CLINICAL TRIAL: NCT04354402
Title: Follow-Up Study of Phase III Study of SyB L-0501 in Combination With Rituximab to Treat Recurrent/Relapsed Diffuse Large B-Cell Lymphoma (Protocol Number: 2017002)
Brief Title: Follow-up Study of SyB L-0501 in Combination With Rituximab to Treat DLBCL
Status: Completed | Type: Observational
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019001
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study is a follow-up study to update the survival time data (overall survival, progression-free survival, and duration of response) of the subjects who received SyB L-0501 at least once in Phase III Study of SyB L-0501 in combination with rituximab to treat recurrent/relapsed diffuse large B-cell lymphoma study (2017002) by reviewing their follow-up information following the study completion of Study 2017002.

In this study, the follow-up information gathered until the end of the investigation period is reviewed after obtaining informed consent from the subjects or their legal representatives. Accordingly, no intervention, such as administration of the investigational product or examination, will be performed.

Investigative methods

1. The investigator or subinvestigator gives an explanation to a subject or his/her legal representative to obtain written informed consent to provision of information pertaining to this study.
2. After obtaining informed consent, the investigator or subinvestigator reviews the follow-up information following the completion of Study 2017002 in source documents regarding the following items:

1. Survival status 2. Aggravation (progression or recurrence) 3. Drugs or procedures used for treatment of DLBCL or prophylaxis against its progression or recurrence 4. Occurrence of other malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who received the investigational product at least once in Study 2017002
2. Subjects who or whose legal representatives gave written informed consent to provision of data pertaining to this study

Exclusion Criteria:

1. Subjects whose death was confirmed during the outcome investigation period in Study 2017002

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects who received SyB L-0501 at least once in Phase III Study of SyB L-0501 in combination with rituximab to treat recurrent/relapsed diffuse large B-cell lymphoma study (2017002) and who (or their legal representatives) give informed consent.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 8 months
  The length of time from the date of case registration in Study 2017002 to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 8 months
  The length of time from the date of treatment initiation (Day 1) in the first cycle in Study 2017002 to the date of progression (including recurrence/relapse), death from any cause, or censoring.
Duration of Response (DOR) | Up to 8 months
  The length of time from the date when complete response (CR) or partial response (PR) was achieved in Study 2017002 to the date of progression (including recurrence/relapse), death from any cause, or censoring.

CONTACTS AND LOCATIONS:
Locations (17):
- Japan (17):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Matsuyama, Ehime
  - Research Site, Ōta, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sayama, Osaka
  - Research Site, Izumo, Shimane
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Koto, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Akita
  - Research Site, Fukuoka
  - Research Site, Ibaraki
  - Research Site, Kyoto
  - Research Site, Nagasaki
  - Research Site, Osaka
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Murayama K, Kiguchi T, Izutsu K, Kameoka Y, Hidaka M, Kato H, Rai S, Kuroda J, Ishizawa K, Ichikawa S, Ando K, Ogura M, Fukushima K, Terui Y. Bendamustine plus rituximab in Japanese patients with relapsed or refractory diffuse large B-cell lymphoma. Ann Hematol. 2022 May;101(5):979-989. doi: 10.1007/s00277-022-04801-2. Epub 2022 Mar 4. PMID 35244756